CLINICAL TRIAL: NCT02098317
Title: Efficacy and Tolerability of Vitamin D and Docosahexaenoic Acid (DHA) in Children With Biopsy Proven NAFLD
Brief Title: DHA and Vitamin D in Children With Biopsy-proven NAFLD
Acronym: VitD_DHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Professor, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VD3_DHA_NAFLD
Record Dates: First submitted 2014-03-24; First posted 2014-03-28 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: NAFLD; Non Alcoholic Steatohepatitis (NASH)
Keywords: NAFLD; NASH; DHA; VITAMIN D; OBESITY; CHILDREN
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- TREATED GROUP (Experimental): this group will treated with pearls containing DHA plus Vitamin D3 (500 mg and 800 IU, respectively) given orally in association with lifestyle intervention [hypocaloric diet (25-30 Kcal/kg/day) or isocaloric (40-45 Kcal/kg/day) and physical activity] for 24 weeks
  Interventions: Drug: DHA plus Vitamin D
- PLACEBO GROUP (Placebo Comparator): this group will treated with identical placebo pearls given orally in association with lifestyle intervention [hypocaloric diet (25-30 Kcal/kg/day) or isocaloric (40-45 Kcal/kg/day) and physical activity] for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHA plus Vitamin D — DHA 500 mg plus Vitamin D 800 IU
  Arms: TREATED GROUP
Drug: Placebo — Placebo pearls mimicking pearls with DHA and Vitamin D
  Arms: PLACEBO GROUP

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has reached epidemic proportions and is rapidly becoming the one of most common causes of chronic liver disease in children. The pathogenesis of NAFLD is generally considered the result of a series of liver injuries, commonly referred as "multi-hit" hypothesis. Several studies suggest that inflammatory pathways and oxidative stress could be responsible of disease progression.

The purpose of this interventional study is to evaluate the efficacy and tolerability of docosahexaenoic acid (DHA) and Vitamin D in children and adolescents with biopsy-proven nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Sixty-six children or adolescents (4-16 years) with liver biopsy proven NAFLD will be enrolled. They will be randomized to treatment with DHA and Vitamin D (n=33) or an identical placebo (n=33) given orally for a period of 6 months. All patients will be included in a lifestyle intervention program consisting of a diet tailored on the individual requirements and physical exercise.

Patients will undergo a medical evaluation at 3-6 and 12 months during the 12-months study period. Liver biopsy will be performed at baseline and at 12 months. Anthropometric measurements and laboratory tests, including liver enzymes, gluco-insulinemic profile and lipids will be performed at baseline and repeated at 6-12 months

ELIGIBILITY:
Inclusion Criteria:

* biopsy consistent with the diagnosis of NAFLD/NASH
* reduced serum levels of vitamin D aminotransferases (ALT) levels <10 upper limit of normal
* hyperechogenicity at liver ultrasound examination suggestive of fatty liver
* International normalized ratio (INR) < 1,3
* Albumin > 3 g/dl
* total bilirubin < 2,5 mg/dl
* no previous gastrointestinal bleeding
* no previous portosystemic encephalopathy
* normal renal function
* no hepatitis B, hepatitis C infection
* normal cell blood count

Exclusion Criteria:

* alcohol consumption
* use of drugs known to induce steatosis or to affect body weight and carbohydrate metabolism
* autoimmune liver disease, metabolic liver disease, Wilson's disease, and a-1-antitrypsin-associated liver disease
* every clinical or psychiatric disease interfering with experimentation according to investigator's evaluation
* finding of active liver disease due to other causes

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement in NAFLD Activity Score (NAS) | 12 months

SECONDARY OUTCOMES:
improvement of laboratory parameters of metabolic syndrome, such as lipids and gluco-insulinemic profile | at 6 and 12 months
safety | 6 months
  clinical examination, medical history and specific laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, Professor, Principal Investigator — Bambino Gesù Children Hospital
Locations (1):
- Bambino Gesù Children Hospital, Rome, Italy, Italy